CLINICAL TRIAL: NCT05051956
Title: Evaluation of the G8 Questionnaire and the Groningen Frailty Indicator to Predict Toxicities of CDK 4/6 Inhibitors in Older Breast Cancer Patients?
Brief Title: Evaluation of Geriatric Questionnaires to Predict Toxicities of CDK 4/6 Inhibitors in Older Breast Cancer Patients?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Asoc. Prof. Erdoğan Selçuk Şeber, Assoc. Prof., Namik Kemal University
Other Study IDs: Geriatric-CDK4/6
Record Dates: First submitted 2021-09-15; First posted 2021-09-21 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Can the Geriatric Questionnaires Predict Adverse Effects in Geriatric Breast Cancer Patients Treated With Cyclin-dependent Kinase 4 and 6 Inhibitors
MeSH Terms: interventions — palbociclib; ribociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CDK4/6 inhibitors: The patient who is started on one of the CDK 4/6 inhibitors (palbociclib 125 mg 3 weeks on 1 week off) or ribociclib 600 mg 3 weeks on 1 week off) will be followed up for adverse events.
  Interventions: Drug: Palbociclib 125mg and Ribociclib 600 mg

INTERVENTIONS:
Drug: Palbociclib 125mg and Ribociclib 600 mg — Administration of Palbociclib or Ribociclib

SUMMARY:
CDK 4/6 inhibitors (palbociclib, ribociclib) have taken their place in our practice recently with their clinical benefits in the treatment of hormone-positive and HER2 negative metastatic breast cancer. Abemaciclib, another CDK 4/6 inhibitor, is not frequently preferred because of reimbursement problems in Turkey. The most obvious advantages of CDK 4/6 inhibitors are that they are used orally and have relatively fewer side effects against chemotherapy. Neutropenia, diarrhea, elevation in liver function tests are the main dose-limiting side effects. In the geriatric age group, it can be thought that the expected benefit from the treatment will not be achieved in cases where these side effects cannot be predicted or managed well. The geriatric age group (65 years and older) deserves special attention in oncology practice, considering both the treatments and the disease itself. Although a number of very useful clinical scales have been developed regarding this subject, it is important that the scale used should be comprehensive as well as being easily applicable for integrating it into daily practice. Geriatric 8 (G8) was found to be a highly sensitive test based on a comprehensive geriatric examination, while the Groningen frailty scale with high specificity. The common feature of these two tests is that they are suitable for daily practice as they are easy to fill. In the light of this information, we aimed to examine whether the G8 and Groningen frailty scale could shed light on clinicians in predicting side effects during the use of CDK 4/6 inhibitors (palbociclib and ribociclib) in geriatric breast cancer patients. We also aimed to reveal the adverse events of these CDK 4/6 inhibitors as real-life experience.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer 65 years and older Treated with CDK 4/6 inhibitors (Palbociclib or Ribociclib)

Exclusion Criteria:

* Below 65 years old

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric (65 years and older) breast cancer patients treated with CDK4/6 inhibitors (Palbociclib or Ribociclib)
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Adverse Event | 6 months period
  First and second adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Birol Ocak, MD, Principal Investigator — Uludag University; Özlem Aydın İsak, MD, Principal Investigator — Ankara Dışkapı Yıldırım Beyazıd Training and Research Hospital; Elif Şenocak Taşçı, MD, Principal Investigator — Mehmet Ali Aydınlar Acıbadem University; Seher Yıldız Tacar, MD, Principal Investigator — Dr. Sadi Konuk Bakırköy Training and Research Hospital; Müslih Ürün, MD, Principal Investigator — Eskişehir City Hospital; Sema Türker, MD, Principal Investigator — Zonguldak Atatürk Public Hospital; Turgut Kaçan, Assoc. Prof, Principal Investigator — Bursa Yüksek İhtisas Training and Research Hospital; Özlem Özdemir, MD, Principal Investigator — İzmir Bozyaka Training and Research Hospital; Eda Tanrıkulu Şimşek, MD, Principal Investigator — Haydarpaşa Numune Training and Research Hospital; Hasan Çağrı Yıldırım, MD, Principal Investigator — Hacettepe University; Teoman Şakalar, MD, Principal Investigator — Kahramanmaraş Necip Fazıl City Hospital; Gülhan İpek Deniz, MD, Principal Investigator — Private Tansan Clinic; Mustafa Ersoy, MD, Principal Investigator — Eskişehir Osmangazi University; Yusuf Karakaş, MD, Principal Investigator — Acıbadem Bodrum Hospital; Ezgi Değerli, MD, Principal Investigator — İstanbul University Cerrahpaşa Medicine Faculty; Hacer Demir, MD, Principal Investigator — Afyon University of Health Sciences; Sinem Akbaş, MD, Principal Investigator — Koç University Hospital; Ahmet Gülmez, MD, Principal Investigator — İnönü University; Özkan Alan, Assoc. Prof., Principal Investigator — Tekirdağ Fehmi Cumalıoğlu City Hospital; Rukiye Arıkan, MD, Principal Investigator — Marmara University; Özden Özer, MD, Principal Investigator — Dokuz Eylul University; Sercan Ön, MD, Principal Investigator — Ege University; Zahid Koçak, MD, Principal Investigator — Necmettin Erbakan University; Nil Molinas Mandel, Prof., Principal Investigator — Koç University; Onur Eşbah, Prof., Principal Investigator — Duzce University; Ali İnal, Assoc. Prof., Principal Investigator — Mersin City Hospital; Murat Araz, Assoc. Prof., Principal Investigator — Necmettin Erbakan University; Halil Taşkaynatan, MD, Principal Investigator — İzmir Private Ege City Hospital; Abdullah Sakin, Assoc. Prof., Principal Investigator — Yuzuncu Yil University; Eyyüp Çavdar, MD, Principal Investigator — Namik Kemal University; Kubilay Karaboyun, MD, Principal Investigator — Namik Kemal University; Erdoğan Selçuk Şeber, Assoc. Prof., Principal Investigator — Namik Kemal University
Locations (1):
- Tekirdağ Namık Kemal University, Tekirdağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No